CLINICAL TRIAL: NCT03655574
Title: Brief Individual and Parent Interventions for Substance Use in Truant Adolescents
Brief Title: Substance Use Interventions for Truant Adolescents
Acronym: GOALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1802001993; 1R01DA045396-01A1 (NIH)
Record Dates: First submitted 2018-08-01; First posted 2018-08-31 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Adolescent Problem Behavior; Truancy; Unsocialized; Marijuana Abuse; Truancy; Socialized; Substance Abuse; Alcohol Abuse
Keywords: Brief intervention; Behavioral intervention; Juvenile justice; Motivational enhancement
MeSH Terms: conditions — Marijuana Abuse; Substance-Related Disorders; Alcoholism

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be informed about which intervention arm they receive. Assessors will have the condition of the participant masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational + Family Check-up (MET+FCU) (Experimental): The MET individual session covers three constructs; 1) intentions to use marijuana; 2) normative beliefs about peer substance use; and 3) attitudes towards peer substance use. These same three constructs are also addressed with respect to truancy. In addition, motivation to abstain from substance use is discussed.
  The FCU session with teens and parents/caregivers begins by collecting self-report measures and conducting a videotaped Family Assessment Task (FAsTask) to assess parent-teen interactions. The FAsTask is the basis of FCU feedback. There are four specific phases of the feedback session: 1) Self-assessment, 2) Support and clarification, 3) Feedback, and, 4) Action plan.
  Interventions: Behavioral: Motivational + Family Check-up (MET+FCU)
- Psychoeducation (Placebo Comparator): An interventionist will review a set of educational materials with the parents regarding teen marijuana use, effects of marijuana on the brain, body and behavior, risks associated with marijuana use, how to tell if a teen is engaging in marijuana use or truancy, and parenting skills. A comparable set of materials will be reviewed with the adolescent.
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Behavioral: Motivational + Family Check-up (MET+FCU) — In the MET session, motivational strategies of individualized normative feedback, examining decisional balance, and providing information/advice will be used to support goals for behavior change and to examine barriers to changes. There are four specific phases of the FCU session: (1) Self-assessment: Parents are asked if they learned anything about their family from participating in the assessment. (2) Support and clarification: The interviewer supports the parent's self-assessment efforts, assesses their level of understanding, and clarifies issues within the family. (3) Feedback: A summary form of the assessment is reviewed. (4) Action Plan: Throughout the session, the counselor works with the parent to develop a brief, written Action Plan about communication and monitoring.
  Arms: Motivational + Family Check-up (MET+FCU)
Other: Psychoeducation — Psychoeducation about substances is provided to teens and parents.
  Arms: Psychoeducation

SUMMARY:
This study evaluates a brief motivation-building intervention for parents and teens to reduce truancy and substance use. It is hypothesized that the motivational intervention will result in better outcomes compared to an education-only intervention.

DETAILED DESCRIPTION:
Adolescents who use marijuana and are truant from school are a high-risk population with increased likelihood of substance use disorders, criminal justice involvement, and long-term impairments in vocational, family, and peer domains.

This study will test a theory-driven intervention for early adolescent marijuana using, truant youth identified through Rhode Island Truancy and Family Courts. Adolescents will be randomly assigned to one of the 2 conditions: a motivational interview versus psychoeducation.

ELIGIBILITY:
Inclusion Criteria:

* the target child is in 6th-10th grade at the start of the project and living at home with at least one parent/guardian,
* the teen must report 6 or more incidences of marijuana use in the last 90 days (an approximation of biweekly use)
* by law, the teen must have at least 20 unexcused absences in an academic year to be in truancy court, and (4) parental consent and teen assent are obtained.

Exclusion Criteria:

* the family is not able to speak and understand English or Spanish well enough to complete study procedures
* developmental delay, as determined by school placements outside the regular classroom, that would affect comprehension of the intervention.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Frequency of Marijuana Use | Last 90 days at baseline, and 3, 6, and 12 months
  Total number of marijuana use days .
Change in Quantity of Marijuana Use per Occasion of Use | Last 90 days at baseline and 3, 6, and 12 months
  Average quantity of marijuana use per day

SECONDARY OUTCOMES:
Change in Days truant from school | Last 90 days at baseline, and 3, 6, and 12 months
  School attendance based on objective school records
Change in Days truant from school, self-report | Last 90 days at baseline, and 3, 6, and 12 months
  School attendance based on self-report

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Spirito, Ph.D., Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Rhode Island Family Court, Providence, Rhode Island
  - Brown Univerity, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
The final study protocol will contain the information necessary to reproduce the findings in other populations. The protocol will include a copy of this grant application including Specific Aims and study population; recruitment and enrollment information; the measures collected and coding of the measures and subscales; the clinician intervention procedures; data analyses; syntax for data summary, and data analysis plans
Supporting Information: Study Protocol, SAP, ICF
Time Frame: I year after completion of all data collection
Access Criteria: Contact PI

DOCUMENTS (1):
  • Informed Consent Form (2020-02-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT03655574/ICF_000.pdf